CLINICAL TRIAL: NCT00122980
Title: Stroke With Transfusions Changing to Hydroxyurea
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study has been stopped due to safety and futility concerns.
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SWiTCH; 1U01HL078787-01A1 (NIH)
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-08

CONDITIONS: Hemochromatosis; Cerebrovascular Accident; Anemia, Sickle Cell; Hematologic Diseases
Keywords: Blood Diseases
MeSH Terms: conditions — Hemochromatosis; Stroke; Anemia, Sickle Cell; Hematologic Diseases | interventions — Erythrocyte Transfusion; Iron Chelating Agents; Hydroxyurea; Phlebotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Hydroxyurea and phlebotomy
  Interventions: Drug: Hydroxyurea; Procedure: Phlebotomy
- 2 (Active Comparator): Transfusion and chelation
  Interventions: Procedure: Red Cell Transfusions; Procedure: Iron Chelation

INTERVENTIONS:
Procedure: Red Cell Transfusions — Red Blood Cell Transfusions
  Arms: 2
Procedure: Iron Chelation — Iron Chelation Therapy
  Arms: 2
Drug: Hydroxyurea — Hydroxyurea
  Arms: 1
Procedure: Phlebotomy — Phlebotomy
  Arms: 1

SUMMARY:
The purpose of this study is to compare standard therapy (transfusions and chelation) with alternative therapy (hydroxyurea and phlebotomy) for the prevention of secondary stroke and management of iron overload in children with sickle cell anemia (SCA).

DETAILED DESCRIPTION:
BACKGROUND:

Stroke occurs in 10% of children with SCA and has a very high risk of recurrence without therapy. Affected children receive chronic erythrocyte transfusions to prevent a secondary stroke, which are effective but have limited long-term utility due to transmission of infectious agents, erythrocyte alloantibody and autoantibody formation, and iron overload. Transfusion acquired iron overload can cause chronic organ damage with hepatic fibrosis and cirrhosis, poor growth and development, cardiac arrhythmias, and early sudden death in young patients with SCA and stroke. An alternative to transfusions for secondary stroke prevention that also addresses the issue of transfusion acquired iron overload is clearly needed. Hydroxyurea can prevent acute vaso-occlusive events in SCA, but its utility for cerebrovascular disease and for the prevention of secondary stroke in SCA is not proven. Pilot data indicate hydroxyurea can prevent stroke recurrence in children with SCA; after transfusions are discontinued, serial phlebotomy reduces iron burden.

DESIGN NARRATIVE:

This is a Phase III randomized clinical trial for children with SCA. The hypothesis is that hydroxyurea and phlebotomy can maintain an acceptable stroke recurrence rate and significantly reduce the hepatic iron burden. The primary aim is to compare standard therapy (transfusions and chelation) with alternative therapy (hydroxyurea and phlebotomy) for the prevention of secondary stroke and management of iron overload. Additional aims include comparisons of growth and development, frequency of non-stroke neurological and other sickle-related events, and quality of life. The use of hydroxyurea for secondary stroke prevention, coupled with removal of excess iron by phlebotomy, would represent a significant improvement in the management of individuals with SCA and stroke. If hydroxyurea is effective for the prevention of secondary stroke, it may also be beneficial for other children with SCA and cerebrovascular disease, including those at risk for primary stroke.

The trial includes approximately 130 children (5.0-18.9 years of age with 65 subjects per treatment arm) with SCA who have had symptomatic cerebral infarctions and have been treated with red cell transfusions for at least 18 months. After completing baseline screening studies, half the participants will be switched to a therapeutic program of hydroxyurea and phlebotomy. Half of the participants will remain on transfusion and chelation. The composite primary endpoint in this study is to compare two modalities of treatment for the prevention of secondary stroke and management of iron overload. The impetus for this trial is the fact that long-term transfusion and chelation therapy in children is difficult, is frequently unsuccessful, and is often complicated by severe symptomatic iron overload, particularly of the heart, lungs, and liver.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects with severe forms of sickle cell anemia (HbSS, HbSβ0 thalassemia, HbSOArab)
* Age range of 5.0-18.9 years, inclusive, at the time of study entry
* Initial (primary) completed overt clinical stroke after the age of one year (12 months) with documented infarction on brain computed tomography (CT) or magnetic resonance imaging (MRI)
* At least 18 months of chronic monthly erythrocyte transfusions since primary stroke
* Transfusional iron overload, defined as a previously documented liver iron concentration (LIC) greater than or equal to 5.0 mg Fe per gram of dry weight liver or serum ferritin greater than or equal to 500 ng/mL on two independent measurements
* Adequate monthly erythrocyte transfusions with average HbS less than or equal to 45% (the upper limit of the established academic community standard) in the 6 months prior to study entry
* Parent or guardian willing and able to provide informed consent with verbal or written assent from the child (less than 18 years of age) or subject willing and able to provide informed consent (older than 18 years of age)
* Ability to comply with study-related treatments, evaluations, and follow-up

Exclusion Criteria:

* Inability to receive or tolerate chronic red blood cell (RBC) transfusion therapy, due to any of the following:

  1. Multiple RBC alloantibodies making cross-matching difficult or impossible
  2. RBC autoantibodies making cross-matching difficult or impossible
  3. Religious objection to transfusions that preclude their chronic use
  4. Non-compliance with transfusions in the 6 months prior to study entry (temporary exclusion)
* Inability to take or tolerate daily oral hydroxyurea, due to any of the following:

  1. Known allergy to hydroxyurea therapy
  2. HIV infection
  3. Cancer
  4. Pregnant or breastfeeding
  5. Previous stem cell transplant or other myelosuppressive therapy
* Clinical and laboratory evidence of hypersplenism, due to any of the following:

  1. Palpable splenomegaly greater than 5 cm below the left costal margin and
  2. Transfusion requirement greater than 250 mL/kg in the 12 months prior to study entry
* Abnormal laboratory values at initial evaluation (temporary exclusion):

  1. Pre-transfusion hemoglobin concentration less than 7.0 gm/dL
  2. White blood cell (WBC) count less than 3.0 x 109/L
  3. Absolute neutrophil count (ANC) less than 1.5 x 109/L
  4. Platelet count less than 100 x 109/L
  5. Serum creatinine more than twice the upper limit for age OR greater than or equal to 1.0 mg/dL
* Current participation in other therapeutic clinical trials
* Current use of other therapeutic agents for SCA (e.g., arginine, decitabine, magnesium)
* Any condition or chronic illness, such as a positive tuberculin (PPD) test, which in the opinion of the study physician makes study participation ill-advised
* Inability or unwillingness to complete required screening studies, including blood tests, brain MRI/magnetic resonance angiography (MRA), and liver biopsy
* A sibling enrolled in SWiTCH

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 134 (Actual)
Dates: Start 2006-10; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell E. Ware, MD, PhD, Principal Investigator — Baylor College of Medicine; Ronald W. Helms, PhD, Principal Investigator — Rho Incorporated
Locations (28):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami, Jackson Memorial Hospital, Miami, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Grady, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Wayne State University, Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Children's Mercy Hospital, Kansas City, Missouri
  - St. Joseph's Children's Hospital, Paterson, New Jersey
  - State University of New York/Downstate Medical Center, Brooklyn, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Columbia University Medical Center, Morgan Stanley Children's Hospital of New York-Presbyterian, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - East Carolina University, Greenville, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Helton KJ, Adams RJ, Kesler KL, Lockhart A, Aygun B, Driscoll C, Heeney MM, Jackson SM, Krishnamurti L, Miller ST, Sarnaik SA, Schultz WH, Ware RE; SWiTCH Investigators. Magnetic resonance imaging/angiography and transcranial Doppler velocities in sickle cell anemia: results from the SWiTCH trial. Blood. 2014 Aug 7;124(6):891-8. doi: 10.1182/blood-2013-12-545186. Epub 2014 Jun 9. PMID 24914136
- [Derived] Alvarez O, Yovetich NA, Scott JP, Owen W, Miller ST, Schultz W, Lockhart A, Aygun B, Flanagan J, Bonner M, Mueller BU, Ware RE; Investigators of the Stroke With Transfusions Changing to Hydroxyurea Clinical Trial (SWiTCH). Pain and other non-neurological adverse events in children with sickle cell anemia and previous stroke who received hydroxyurea and phlebotomy or chronic transfusions and chelation: results from the SWiTCH clinical trial. Am J Hematol. 2013 Nov;88(11):932-8. doi: 10.1002/ajh.23547. Epub 2013 Aug 30. PMID 23861242
- [Derived] Ware RE, Helms RW; SWiTCH Investigators. Stroke With Transfusions Changing to Hydroxyurea (SWiTCH). Blood. 2012 Apr 26;119(17):3925-32. doi: 10.1182/blood-2011-11-392340. Epub 2012 Feb 7. PMID 22318199
- [Derived] Ware RE, Schultz WH, Yovetich N, Mortier NA, Alvarez O, Hilliard L, Iyer RV, Miller ST, Rogers ZR, Scott JP, Waclawiw M, Helms RW. Stroke With Transfusions Changing to Hydroxyurea (SWiTCH): a phase III randomized clinical trial for treatment of children with sickle cell anemia, stroke, and iron overload. Pediatr Blood Cancer. 2011 Dec 1;57(6):1011-7. doi: 10.1002/pbc.23145. Epub 2011 Aug 8. PMID 21826782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III First Patient In: 31-October-2006; Last Patient Last Visit: 15-December-2010; 25 medical clinics in the United States of America.
Pre-assignment Details: Participant qualification was initially evaluated by medical chart review and interview. Subsequent to subject consent, subjects were further screened to confirm eligibility. Screening included, in part, expert verification of initial stroke and of liver biopsy results prior to randomization.
Groups:
- Hydroxyurea/Phlebotomy: 1: The Hydroxyurea/Phlebotomy group includes participants randomized to Alternative Treatment. Participants commenced hydroxyurea treatment at 20 mg/kg/day with step-wise escalation to maximum tolerated dose (MTD) defined by mild myelosuppression (absolute neutrophil count 2-4 x 10^9/L). Transfusions continued for 4-9 months during an overlap phase using a modified schedule to protect against recurrent stroke during hydroxyurea dose escalation. Once MTD was reached and transfusions were discontinued, phlebotomy commenced with a target of 10 mL/kg (maximum volume 500mL) blood removed monthly to reduce iron burden. Lower phlebotomy volumes (5 mL/kg) were recommended if participants were excessively anemic (hemoglobin concentration 7.0-7.9 gm/dL); phlebotomy was not performed if the hemoglobin level was <7.0 gm/dL. The total duration of study treatment was 30 months after randomization, with a final study visit scheduled 6-months after discontinuation of study treatments.
- Transfusion/Chelation: 2: The Transfusion/Chelation group includes participants randomized to Standard Treatment. Participants continued to receive monthly blood transfusions designed to maintain ≤30% HbS, with local discretion regarding type of transfusion (e.g., simple or erythrocytapheresis). These participants also received daily iron chelation typically with deferasirox (Exjade®). Children already on chelation initially maintained their current dose, while those starting deferasirox received 20 mg/kg/day, with dose escalation in both groups as indicated and tolerated.
Period: Overall Study
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation
Started | 67 (Randomized sample: 67; Intent-to-treat sample: 67) | 66 (Randomized sample: 67; Intent-to-treat sample: 66)
Completed | 24 (Study terminated early) | 26 (Study terminated early)
Not Completed | 43 | 40
Not completed — Death | 0 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 5 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Adjudicated stroke (study endpoint) | 7 | 0
Not completed — Study termination | 27 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation | Total
Number analyzed (Participants) | 67 | 66 | 133
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60 | 60 | 120
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 13.0 (4.05) | 13.3 (3.76) | 13.1 (3.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 35 | 61
  Male | 41 | 31 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 63 | 64 | 127
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — NIH race categories
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 62 | 64 | 126
    White | 0 | 0 | 0
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 67 | 66 | 133
History of splenomegaly [Number; unit: Participants] — History of Splenomegaly is defined as participants who ever were diagnosed with splenomegaly. Splenomegaly includes hypersplenism (enlarged spleen with platelet count < 150 x 10^9/L), splenic sequestration (enlarged spleen with decrease in steady state hemoglobin of at least 2 gm/dL and/or platelet count < 150 x 10^9/L), and/or Splenomegaly without hypersplenism. Repeated dose-limiting toxicities may reflect the development of splenomegaly and hypersplenism. The size of the spleen was assessed monthly during the study
  Participants
    Yes | 22 | 16 | 38
    No | 45 | 50 | 95
Age at index stroke [Mean (Standard Deviation); unit: years] — Index Stroke is defined as an overt clinical stroke after the age of one year (12 months) with documented infarction on brain computed tomography (CT) or MRI.
  years | 5.6 (2.97) | 6.2 (2.75) | 5.9 (2.87)
Duration of Transfusion [Mean (Standard Deviation); unit: years] — Duration of Transfusions refers to the duration of chronic transfusion therapy (either simple, partial exchange, or erythrocytapheresis)for secondary stroke prevention.
  years | 7.4 (3.85) | 7.0 (3.61) | 7.2 (3.72)
Prior use of Desferal (deferoxamine mesylate) [Number; unit: participants] — Desferal (deferoxamine mesylate) is a chelation therapy to reduce hepatic iron overload and was used in a subset of the Transfusion/Chelation treatment group of this study.
  participants
    Yes | 47 | 44 | 91
    No | 19 | 19 | 38
    Missing | 1 | 3 | 4
Prior use of Exjade (deferasirox) [Number; unit: participants] — Exjade (deferasirox) is a chelation treatment to reduce hepatic iron overload and was used in a subset of the Transfusion/Chelation treatment group of this study.
  participants
    Yes | 57 | 55 | 112
    No | 9 | 8 | 17
    Missing | 1 | 3 | 4
Prior use of hydroxyruea [Number; unit: participants] — Hydroxyurea, in combination with phlebotomy, is the Alternative Treatment to prevent secondary stroke in this study.
  participants
    Yes | 5 | 3 | 8
    No | 62 | 63 | 125
Liver iron concentration [Median (Inter-Quartile Range); unit: mg ferritin/gram dry weight liver] — Participants were included in this trial if they had transfusional iron overload, defined as previously documented liver iron concentrations (LIC) ≥5.0 mg Fe per gram of dry weight liver or serum ferritin ≥500 ng/mL on 2 independent measurements. Part of the composite primary endpoint hypothesis of this study is that liver iron levels will decrease more in the Hydroxyurea/Phlebotomy group than in the Transfusion/Chelation group.
  mg ferritin/gram dry weight liver | 14.5 [9.5 to 23.3] | 13.9 [8.7 to 22.9] | 14.5 [9.0 to 23.0]
History of recurrent stroke [Number; unit: participants] — Recurrent stroke at baseline is defined as having had more than one stroke prior to study entry.
  participants
    Yes | 10 | 4 | 14
    No | 57 | 62 | 119

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of an Adjudicated Secondary Stroke During the 30-month Treatment Period
Description: Secondary stroke is the first component of the composite primary endpoint and considers the number of participants with recurrent secondary stroke events during 30 months of treatment. Stroke was defined as any clinical event with brain injury due to vascular disease. All neurological events underwent formal stroke adjudication.
Time Frame: Because the study was terminated early, time frame is from beginning of treatment until end of treatment (up to 30 Months)
Population: The Intent-to-Treat population included all subjects who were randomized and who received any on-study treatment.
Measure: Number; unit: participants
Groups:
- Hydroxyurea/Phlebotomy: Hydroxyurea and Phlebotomy Group (Alternative Treatment Arm)
- Transfusion/Chelation: Transfusion and Chelation Group (Standard Treatment Arm)
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation
Number analyzed (Participants) | 67 | 66
participants
  Stroke | 7 | 0
  No Stroke | 60 | 66
Statistical Analysis 1: Comparison: Hydroxyurea/Phlebotomy vs Transfusion/Chelation; Concluding that Hydroxyurea/Phlebotomy group is better than the Transfusion/Chelation group required rejecting the STROKE null hypothesis in favor of the alternative: Hydroxyurea/Phlebotomy recurrent stroke rate is less than Transfusion/Chelation rate plus 0.20, the non-inferiority margin, AND rejecting the IRON null hypothesis in favor of the alternative: Hydroxyurea/Phlebotomy baseline-adjusted mean LIC is less than for Transfusion/Chelation (see next primary endpoint analysis); Test type: Non-Inferiority or Equivalence — Based on pilot data, the efficacy of hydroxyurea to reduce secondary stroke rate was not predicted to be equivalent to transfusions. Therefore, an increased stroke rate (non-inferiority margin = 0.20) was allowed by study design. This "acceptable" stroke margin was predicted to be offset by the likelihood of significantly greater improvement in the management of iron overload through elimination of transfusions along with serial phlebotomy in the Hydroxyurea/Phlebotomy arm; p = 0.214, Log Rank

2. Primary Outcome: Liver Iron Content (LIC) Change-from-baseline
Description: LIC change-from-baseline is the second component of the composite primary endpoint. LIC was measured by quantitative liver biopsy at baseline and at 30 months or exit from the study.LIC values were transformed into Log10 values prior to computing the change from baseline.
Time Frame: as for outcome 1
Population: Intent-to-treat AND both baseline and 30-month post-treatment LICs.
Measure: Log Mean (Standard Deviation); unit: mg ferritin/gram dry weight liver
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation
Number analyzed (Participants) | 31 | 25
mg ferritin/gram dry weight liver | -0.006 (0.187) | -0.120 (0.387)
Statistical Analysis 1: Comparison: Hydroxyurea/Phlebotomy vs Transfusion/Chelation; Concluding that Hydroxyurea/Phlebotomy group is better than the Transfusion/Chelation group required rejecting the STROKE null hypothesis (see previous primary endpoint analysis) in favor of the alternative: Hydroxyurea/Phlebotomy recurrent stroke rate is less than Transfusion/Chelation rate plus 0.20 AND rejecting the IRON null hypothesis in favor of the alternative: Hydroxyurea/Phlebotomy baseline-adjusted mean log10 transformed LIC is less than for Transfusion/Chelation; Test type: Superiority or Other; p = 0.144, Mixed Models Analysis — The a priori defined LOCF approach was deemed to be biased due to the study's early termination, and was replaced by this mixed models analysis; Including main effects of age at consent, baseline iron, and treatment group, on observed change from baseline Log10 transformed values only

3. Secondary Outcome: Pediatric Quality of Life (PedsQL) - Parent Report (Change From Baseline)
Description: The PedsQL(TM) Measurement Model is a modular approach to measuring health-related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. It has a Likert 5-points scale (never to almost always) which were transformed to a 0 to 100 scale based on the PedsQL scoring algorithms, higher scores indicating better quality of life characteristics.
Time Frame: Baseline, mid-point (week 64), and study exit after up to 30-month treatment period (due to study termination)
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation
Number analyzed (Participants) | 67 | 66
units on a scale
  Mid-point: Emotional Functioning Score (n=43,54) | -0.99 (19.709) | 5.56 (20.366)
  Exit: Emotional Functioning Score (n=52, 54) | -1.25 (28.265) | 5.65 (27.676)
  Mid-point: Physical Functioning Score (n=43,64) | -1.71 (33.011) | -0.57 (23.195)
  Exit: Physical Functioning Score (n=53, 54) | 2.27 (34.456) | -0.98 (27.884)
  Mid-point: School Functioning (n=43, 54) | 3.14 (23.017) | -3.34 (22.546)
  Exit: School Functioning (n=51,53) | -0.29 (23.074) | 2.83 (24.564)
  Mid-point : Social Functioning Score (n=42, 54) | 3.69 (23.506) | -0.35 (20.858)
  Exit : Social Functioning Score (n=53, 54) | 2.67 (27.679) | -1.11 (27.208)
  Mid-point: Total Functioning Score (n=43, 54) | 0.39 (20.411) | 0.20 (16.974)
  Exit: Total Functioning Score (n=53, 54) | 1.13 (24.391) | 1.09 (20.773)
  Mid-point: Psychosocial Health Summary (n=43,54) | 1.61 (16.574) | 0.59 (17.072)
  Exit: Psychosocial Health Summary (n=53, 54) | 0.33 (21.535) | 2.11 (20.278)
Statistical Analysis 1: Comparison: Hydroxyurea/Phlebotomy vs Transfusion/Chelation; The change-from-baseline scores were analyzed with an analysis of variance model (ANOVA) with treatment as stratum, testing the hypothesis that the average change from baseline scores do not differ between the treatment groups; Test type: Superiority or Other; p > 0.05, ANOVA; The change-from-baseline scores for each scale were analyzed with an analysis of variance model (ANOVA) with treatment as stratum

4. Secondary Outcome: Pediatric Quality of Life (PedsQL) - Child Report (Change From Baseline)
Description: The PedsQLTM Measurement Model is a modular approach to measuring health-related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. It has a Likert 5-points scale (never to almost always) which were transformed to a 0 to 100 scale based on the PedsQL scoring algorithms, higher scores indicating better quality of life characteristics.
Time Frame: Baseline, midpoint (week 64), and study exit (up to 30 months of treatment)
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation
Number analyzed (Participants) | 67 | 66
units on a scale
  Midpoint: Emotional Functioning Score (n=47, 57) | 1.06 (18.236) | 3.51 (22.240)
  Exit: Emotional Functioning Score (n=55, 54) | 3.82 (21.623) | 3.80 (20.022)
  Midpoint: Physical Functioning Score (n=47, 57) | 0.46 (22.642) | 3.18 (16.308)
  Exit: Physical Functioning Score (n=55, 54) | 3.41 (17.639) | 2.03 (20.426)
  Midpoint: School Functioning Score (n=47, 57) | -1.03 (24.437) | 4.56 (21.615)
  Exit: School Functioning Score (n=55, 53) | 1.76 (20.701) | 2.74 (20.418)
  Midpoint: Social Functioning Score (n=46, 57) | 2.39 (19.909) | 1.84 (25.011)
  Exit: Social Functioning Score (n=54, 54) | 3.13 (21.313) | 2.87 (21.732)
  Midpoint: Total Functioning Score (n=47, 57) | 0.35 (16.557) | 3.26 (16.230)
  Exit: Total Functioning Score (n=55, 54) | 2.90 (16.154) | 2.62 (16.593)
  Midpoint: Psychosocial Health Summary (n=47, 57) | 0.28 (17.180) | 3.30 (18.515)
  Exit: Psychosocial Health Summary Score (n=57, 54) | 2.65 (17.278) | 2.93 (16.910)
Statistical Analysis 1: Comparison: Hydroxyurea/Phlebotomy vs Transfusion/Chelation; The change-from-baseline scores were analyzed with an analysis of variance model (ANOVA) with treatment as stratum; Test type: Superiority or Other; p > 0.05, ANOVA; [statistical method as in outcome 3, analysis 1]

5. Secondary Outcome: Barthel Index (Change From Baseline)
Description: The Barthel Index is a measure of activities of daily living (ADL) and assesses the degree of disability in a particular participant. The index records indicators of independence in terms of the disability caused by impairments, such as those that may be sequelae of stroke. The index was used as a record of what the participant did, not as a record of what the participant could do. Barthel scores range from 0 to 100, with higher scores indicating greater independence in daily living activities (caring for oneself).
Time Frame: Baseline and study exit after up to 30-month treatment period (due to study termination)
Population: Intent-to-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation
Number analyzed (Participants) | 67 | 66
units on a scale | -0.33 (4.269) | -0.53 (6.316)
Statistical Analysis 1: Comparison: Hydroxyurea/Phlebotomy vs Transfusion/Chelation; The change-from-baseline to endpoint scores were analyzed with an analysis of variance model (ANOVA) with treatment as stratum; Test type: Superiority or Other; p = 0.841, ANOVA

6. Secondary Outcome: Woodcock-Johnson Test of Cognitive Abilities (WJ-C) and Achievement (WJ-III) (Change From Baseline)-Excluding Verbal
Description: This test is designed to assess both broad and narrow cognitive abilities in children age 4 years and above as well as to measure major aspects of academic achievement in persons aged 2-90 years. Scaled scores range from 0-100. Higher scores mean better abilities/achievements.
Time Frame: Baseline and study exit after up to 30-month treatment period (due to study termination)
Population: Intent-to-Treat. Because the study was terminated, it was not possible to schedule the full battery of neurological assessments on all subjects. Only subjects with both baseline and end of study assessments were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation
Number analyzed (Participants) | 67 | 66
units on a scale
  General intellectual ability (n=33, 35) | -1.64 (9.594) | -3.00 (6.535)
  Processing speed (n=35, 33) | -0.80 (14.046) | 2.06 (13.245)
  Working memory (n=33, 34) | -7.67 (22.545) | -2.65 (9.435)
  Broad attention (n=31, 33) | -4.36 (12.693) | -0.49 (8.220)
  Executive processes (n=32, 33) | -0.72 (9.323) | -1.15 (7.173)
  Broad reading (n=34, 33) | -0.29 (8.615) | -0.94 (5.172)
  Broad math (n=34, 33) | -3.53 (9.542) | -5.76 (14.292)
Statistical Analysis 1: Comparison: Hydroxyurea/Phlebotomy vs Transfusion/Chelation; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p > 0.05, ANOVA

7. Secondary Outcome: Woodcock-Johnson Test of Cognitive Abilities (WJ-C) and Achievement (WJ-III) (Change From Baseline)- Verbal Ability
Description: This test is designed to assess both broad and narrow cognitive abilities in children age 4 years and above as well as to measure major aspects of academic achievement in persons aged 2-90 years. Higher scores mean better abilities/achievements. Scaled scores range from 0-100.
Time Frame: Baseline and study exit after up to 30-month treatment period (due to study termination)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation
Number analyzed (Participants) | 35 | 35
units on a scale | 1.829 (8.305) | -2.487 (8.806)
Statistical Analysis 1: Comparison: Hydroxyurea/Phlebotomy vs Transfusion/Chelation; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.039, ANOVA

8. Secondary Outcome: Growth and Development - Height (Change From Baseline to Endpoint)
Time Frame: Baseline to end of study participation (up to 136 weeks)
Population: Intent-to-Treat with endpoint data
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation
Number analyzed (Participants) | 60 | 60
cm | 4.40 (4.32) | 6.61 (5.87)
Statistical Analysis 1: Comparison: Hydroxyurea/Phlebotomy vs Transfusion/Chelation; Test type: Superiority or Other; p = 0.033, ANCOVA; Analysis controlling for baseline value and time on study

9. Secondary Outcome: Growth and Development - Weight (Change From Baseline to Endpoint)
Time Frame: baseline to end of study participation (up to 136 weeks)
Population: Intent-to-Treat with endpoint data
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation
Number analyzed (Participants) | 64 | 63
kg | 3.83 (5.07) | 6.36 (5.43)
Statistical Analysis 1: Comparison: Hydroxyurea/Phlebotomy vs Transfusion/Chelation; Test type: Superiority or Other; p < 0.01, ANCOVA; Controlling for baseline value and time on study

ADVERSE EVENTS:
Arm/Group | Hydroxyurea/Phlebotomy | Transfusion/Chelation
Serious Adverse Events (participants affected / at risk) | 29/67 | 14/66
Other Adverse Events (participants affected / at risk) | 65/67 | 65/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea/Phlebotomy (N=67) | Transfusion/Chelation (N=66)
Acute chest syndrome (Blood and lymphatic system disorders) | 1 (2) | 3 (3)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 16 (27) | 5 (7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 2 (2)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infusion site infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Near drowning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 6 (7) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Moyamoya disease (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Renal papillary necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea/Phlebotomy (N=67) | Transfusion/Chelation (N=66)
Acute chest syndrome (Blood and lymphatic system disorders) | 6 (7) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 20 (39) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 10 (13) | 1 (1)
Reticulocytopenia (Blood and lymphatic system disorders) | 21 (30) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (9) | 1 (5)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 35 (125) | 29 (75)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 8 (9)
Abdominal pain upper (Gastrointestinal disorders) | 4 (5) | 4 (5)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 12 (15) | 11 (12)
Chest pain (General disorders) | 3 (4) | 4 (4)
Pain (General disorders) | 4 (5) | 5 (5)
Pyrexia (General disorders) | 21 (30) | 20 (37)
Hyperbilirubinaemia (Hepatobiliary disorders) | 9 (22) | 18 (49)
Influenza (Infections and infestations) | 5 (5) | 5 (5)
Sinusitis (Infections and infestations) | 7 (12) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 6 (9) | 5 (6)
Urinary tract infection (Infections and infestations) | 5 (6) | 6 (12)
Viral infection (Infections and infestations) | 6 (6) | 4 (4)
Post procedural complication (Injury, poisoning and procedural complications) | 7 (7) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 4 (4) | 10 (14)
Alanine aminotransferase increased (Investigations) | 15 (25) | 14 (36)
Aspartate aminotransferase increased (Investigations) | 14 (23) | 10 (18)
Blood creatinine increased (Investigations) | 6 (7) | 3 (6)
Transaminases increased (Investigations) | 3 (3) | 5 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (7)
Convulsion (Nervous system disorders) | 2 (8) | 5 (23)
Dizziness (Nervous system disorders) | 5 (5) | 4 (4)
Headache (Nervous system disorders) | 18 (33) | 22 (33)
Transient ischaemic attack (Nervous system disorders) | 3 (4) | 6 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (5)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 8 (11)

LIMITATIONS AND CAVEATS:
The trial was stopped early due to a projected futility of the liver iron component of the primary endpoint in conjunction with the significantly higher number of strokes in the Hydroxyurea/Phlebotomy arm as compared to the Transfusion/Chelation arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No